CLINICAL TRIAL: NCT06040281
Title: The Effects of an Interdisciplinary Treatment Approach in ESRD Patients: a Randomised Controlled Trial
Brief Title: Smart and Fit for Kidney Transplantation
Acronym: S&F4NTx
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: m&i Fachklinik Bad Heilbrunn (Unknown); Carealytix Digital Health GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GE8-2496-IMV-2019-V2
Record Dates: First submitted 2023-09-08; First posted 2023-09-15 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2024-12

CONDITIONS: Chronic Kidney Disease Requiring Chronic Dialysis
Keywords: Transplantation; Prehabilitation; Exercise and Nutritional Support
MeSH Terms: conditions — Motor Activity | interventions — Nutritional Status; Exercise

STUDY DESIGN:
Intervention Model Description: Random assignment in 1:1 ratio to either the intervention group (app-assisted, individual support in nutrition and exercise, three-week comprehensive rehabilitation) or control group (Usual care and app-assisted)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): App-assisted three-week comprehensive rehabilitation individual support in nutrition and exercise
  Interventions: Behavioral: intensive individual support in nutrition and exercise
- Control (Active Comparator): usual care App-assisted
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: intensive individual support in nutrition and exercise — Intensive care for nutrition and exercise adapted to the social context. Individualised exercise and nutrition recommendations.
  three weeks of inpatient rehabilitation with an individual plan of treatment, which includes medical care, sports therapy, physiotherapy, ergotherapy, nutritional education and psychological care App access for comprehensive information about dialysis (nutrition, travel, medication, etc.)
  Arms: Intervention
Behavioral: Usual Care — Usual care App access for comprehensive information about dialysis (nutrition, travel, medication, etc.)
  Arms: Control

SUMMARY:
This study is a randomised controlled intervention trial for patients with chronic kidney disease who are on the waiting list for a kidney transplantation (n=200). The aim of this study is to test the effectiveness of intensive individual nutritional and exercise support combined with comprehensive rehabilitation before transplantation in comparison to a control group.

DETAILED DESCRIPTION:
Patients are randomised to either the intervention or control group at the beginning of the study. Both groups are evaluated at the beginning after 6 months and after 12 months regarding their body composition, physical performance, blood values, quality of life and nutritional status. The control group only receives support via app during the study period (1 year), through which they receive detailed information about dialysis. In addition to access to the app, the intervention group receives individual recommendations for nutrition and exercise as well as a three-week inpatient rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be on dialysis
* Patients ≥ 18 years of age
* Patients who own a smartphone
* Patients must be willing to undergo inpatient rehabilitation within the project period
* signed informed consent and data protection regulation

Exclusion Criteria:

* Patients who are not psychologically or physically able to take part in exercise promotion measures and/or nutritional counselling as well as psychological offers
* Patients who have already participated in a similar project

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-09-18 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
muscle mass | 6 and 12 month
  measured in kg by bio-impedance analysis
body fat mass | 6 and 12 month
  measured in kg by bio-impedance analysis

SECONDARY OUTCOMES:
Six-Minutes-Walk test (6MWT) | 6 and 12 month
  measured in distance (meter)
Sit-to-stand test (STS60) | 6 and 12 month
  measured in number of repetitions in 60 seconds
Timed-up-and-go test (TUG) | 6 and 12 month
  measured in time (seconds)
Quality of life by Short Form Health Survey (SF-12) | 6 and 12 month
  measured in change of scale by questionnaire
Fried Frailty Scale | 6 and 12 month
  measured in change of score (score of 0 = not frail; score of 1-2 = pre-frail; score of 3-5 = frail)
One-Legged Stance Test | 6 and 12 month
  measured in time (seconds)
Stair Climb Test | 6 and 12 month
  measured in time (seconds)

CONTACTS AND LOCATIONS:
Overall Officials: Mario Schiffer, Prof., Study Director — Universitätsklinikum Erlangen
Locations (1):
- Universitätsklinikum Erlangen, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Krusemark H, Kleemann J, Weigand J, Kannenkeril D, Heller K, Hepp T, Albersmeyer M, Gerbig D, Schiffer M. A randomized, controlled, 12-month trial on the effects of an interdisciplinary treatment approach in ESRD patients: study protocol of the smart and fit for kidney transplantation trial (S&F4KTx). Trials. 2025 Aug 21;26(1):298. doi: 10.1186/s13063-025-09022-2. PMID 40841967